CLINICAL TRIAL: NCT03734211
Title: EVOLVD: Cholesterol Lowering With EVOLocumab to Prevent Cardiac Allograft Vasculopathy in De-novo Heart Transplant Recipients
Brief Title: Cholesterol Lowering With EVOLocumab to Prevent Cardiac Allograft Vasculopathy in De-novo Heart Transplant Recipients
Acronym: EVOLVD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lars Gullestad (Other)
Collaborators: Sahlgrenska University Hospital (Other); Skane University Hospital (Other); Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Lars Gullestad, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-005097-19
Record Dates: First submitted 2018-10-26; First posted 2018-11-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Evolocumab; Heart Transplantation; Vasculopathy
MeSH Terms: conditions — Vascular Diseases | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Experimental): Evolocumab (Repatha®) will be administered subcutaneously once monthly in the abdomen, thigh, or upper arm for the duration of the treatment period (one year). The 420 mg evolocumab/placebo will be administered by giving 3 injections consecutively within 30 minutes using the single-use prefilled autoinjector.
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): The placebo is presented in an identical prefilled autoinjector. It is supplied as a sterile, single-use, preservative-free solution for subcutaneous injection in a disposable, spring-based prefilled autoinjector. The prefilled autoinjector contains a 1.0 mL deliverable volume of 1.1% (w/v) sodium carboxymethylcellulose, 250 mM proline, 10 mM acetate, and 0.01% (w/v) polysorbate 80, pH 5.0.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — 420 mg evolocumab will be administered subcutaneously by giving 3 injections consecutively within 30 minutes using the single-use prefilled autoinjector.
  Other Names: Repatha
  Arms: Evolocumab
Drug: Placebo — Placebo will be administered subcutaneously by giving 3 injections consecutively within 30 minutes using the single-use prefilled autoinjector.
  Arms: Placebo

SUMMARY:
The main goal of this study is to evaluate the effect of the proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor evolocumab on cardiac allograft vasculopathy in de novo heart transplant recipients.

Secondary objectives are to assess the impact of treatment on: i) cholesterol levels, ii) renal function, iii) inflammation, iv) quality of life, v) cardiac function as assessed by biomarkers and echocardiography, vi) the number of rejections, and (vii) safety and tolerability. As an exploratory outcome, the investigators will asses the effect of treatment on clinical events (death, myocardial infarction, cerebral stroke, cancer, end stage renal disease).

DETAILED DESCRIPTION:
Cardiac allograft vasculopathy is an important cause of morbidity and mortality in heart transplant recipients. Previous data show that, although clinical coronary artery disease often manifests years after heart transplantation, there are substantial changes in the coronary artery intima thickness over the first year after transplantation, suggesting that the adverse process starts shortly after transplantation. Moreover, the investigator's previous data have suggested that, whereas early intervention can prevent the long-term progression of cardiac allograft vasculopathy, the same intervention is less effective when administered late after heart transplantation. Thus, there seems to be a window of opportunity for preventive measures against cardiac allograft vasculopathy in de-novo transplant recipients.

The strong association between cholesterol levels and coronary heart disease in the general population, the high cholesterol levels in heart transplant recipients, the high prevalence of vasculopathy in the cardiac allograft, and the association between cholesterol levels and cardiac allograft vasculopathy together provide a strong rationale for aggressive cholesterol lowering in heart transplant recipients. Statins improve outcomes in heart transplant recipients, but their limited effect on post-transplant cholesterol levels, adverse effects, and drug interactions contribute to their not providing sufficient prophylaxis against post-transplant atherosclerotic disease.

Evolocumab is a well-tested drug with a favourable safety profile. It effectively reduces cholesterol levels on top of statin therapy in patients with coronary heart disease. The investigators hypothesise that evolocumab on top of statin therapy will significantly lower low density lipoprotein (LDL) levels in de novo heart transplant recipients. The investigators assume that this reduction in cholesterol levels will manifest as a reduced burden of cardiac allograft vasculopathy as measured by intracoronary ultrasound. Ultimately, the investigators believe that a reduced burden of vasculopathy will translate to reduced morbidity and long-term mortality in heart transplant recipients. The EVOLVD trial is a randomised, placebo-controlled, double-blind study designed to test the hypothesis that treatment with evolocumab can ameliorate cardiac allograft vasculopathy in heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Patients will be screened for eligibility during routine follow-up 4 - 8 weeks after heart transplantation. All of the following conditions must apply prior to administering the investigational medicinal product:

* Heart transplant recipient within the last 4 - 8 weeks.
* Age between 18 and 70 years.
* Informed consent obtained and documented according to Good Clinical Practice (GCP), and national/regional regulations.
* No contraindications to coronary angiography with intravascular ultrasound
* Estimated glomerular filtration rate > 20 ml/min/1.73 m2 as assessed by the MDRD formula.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Decompensated liver disease (Child-Pugh class C)
* Severe renal failure, i.e. eGFR < 20 ml/min/1.73 m2 or on renal replacement therapy
* Ongoing rejections or infections
* Known sensitivity or intolerance to evolocumab or any of the excipients of Repatha®
* Prior use of PCSK9 inhibition treatment
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Participation in another clinical trial involving an investigational drug and/or follow-up within 30 days prior to enrolment.
* Pregnancy.
* Female subject who has either (1) not used at least one highly effective method of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment and for an additional 15 weeks after the end of treatment, unless the subject is sterilised or postmenopausal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Maximal intimal thickness | 12 months
  The maximal intimal thickness will be measured by coronary intravascular ultrasound at 12 months after randomization. The maximal intima thickness is defined as the largest distance (in mm) from the intimal leading edge to the external elastic membrane.

SECONDARY OUTCOMES:
Cardiac allograft vasculopathy | 12 months
  Incidence of cardiac allograft vasculopathy, defined as mean a maximal intimal thickness ≥0.5 mm over the entire matched segment, will be measured by intravascular ultrasound 12 months after randomization.
Total atheroma volume | 12 months
  The total atheroma volume will be measured by intravascular ultrasound.
The index of microvascular resistance | 12 months
  The index of microcirculatory resistance will be obtained at the time of routine coronary angiography after heart transplantation at baseline (4-10 weeks) and at the end of treatment 12 months after randomization.
Low-density lipoprotein (LDL) cholesterol | 12 months
  Blood lipids must be assessed after end-of treatment only, to avoid what will effectively amount to study drug allocation unblinding. To avoid bias, the investigators will be blinded to the lipid analyses.
Estimated glomerular filtration rate (eGFR) | 12 months
  The glomerular filtration rate (in in ml/min/1.73 m2) will be estimated by the MDRD formula: 175 x (SCr)-1.154 x (age)-0.203 x 0.742 [if female] x 1.212 [if black], where SCr is serum creatinine in mg/dl, and age is measured in years.
The 36-item short form health survey questionnaire (SF-36) | 12 months
  The SF-36 Health Survey is a 36-item, patient-reported survey of patient health.
The 3-level version of EQ-5D (EQ-5D-3L) questionnaire | 12 months
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
The Beck Depression Inventory (BDI) | 12 months
  The BDI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 12 months
  NT-proBNP values will be used for endpoint analyses.
Cardiac troponin T (TnT) | 12 months
  Troponin T-values will be used for endpoint analyses.
Number of rejections | 12 months
  Number of all rejections will be recorded through the duration of the study.
Number of adverse events (AE) | 12 months
  The standard time period for collecting and recording AE and SAEs will begin at the start of study treatment and will continue for 30 day after end-of treatment (at which time approximately 30 days will have passed since the last study drug injection.
Number of major clinical adverse events | 12 months
  The number of major clinical adverse events, defined as death, myocardial infarction, percutaneous coronary intervention/coronary bypass surgery, cerebral stroke, cancer, end stage renal disease (exploratory endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (5):
- Denmark (2):
  - Department of Cardiology, Rigshospitalet, Copenhagen
  - Department of Cardiology, Aarhus University Hospital, Skejby
- Helsinki University Hospital Heart and Lung Center, Helsinki, Finland
- Sweden (2):
  - Department of Cardiology, Sahlgrenska University Hospital, Gothenburg
  - The Clinic for Heart Failure and Valvular Disease, Skåne University Hospital and Lund University, Lund

REFERENCES:
- [Derived] Broch K, Lemstrom KB, Gustafsson F, Eiskjaer H, Karason K, Gjesdal G, Fagerland MW, Pentikainen M, Lommi J, Gude E, Andreassen AK, Clemmensen TS, Christiansen EH, Bjorkelund E, Berg ES, Arora S, Gullestad L. Randomized Trial of Cholesterol Lowering With Evolocumab for Cardiac Allograft Vasculopathy in Heart Transplant Recipients. JACC Heart Fail. 2024 Oct;12(10):1677-1688. doi: 10.1016/j.jchf.2024.04.026. Epub 2024 Jun 26. PMID 38934968
- [Derived] Broch K, Gude E, Karason K, Dellgren G, Radegran G, Gjesdal G, Gustafsson F, Eiskjaer H, Lommi J, Pentikainen M, Lemstrom KB, Andreassen AK, Gullestad L. Cholesterol lowering with EVOLocumab to prevent cardiac allograft Vasculopathy in De-novo heart transplant recipients: Design of the randomized controlled EVOLVD trial. Clin Transplant. 2020 Sep;34(9):e13984. doi: 10.1111/ctr.13984. Epub 2020 Aug 6. PMID 32445429

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03734211/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03734211/SAP_001.pdf